CLINICAL TRIAL: NCT05772286
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein SOSIP v8.2 763 Vaccine, Adjuvanted With MPLA Liposomes, in Healthy, HIV-Uninfected Adults
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein SOSIP v8.2 763 Vaccine, Adjuvanted With MPLA Liposomes, in Healthy, HIV-Uninfected Adults
Acronym: HIVAC-FOUND
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Polymun Scientific GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-003868-27
Record Dates: First submitted 2023-02-15; First posted 2023-03-16 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 763SIP8/MPLA-5 vaccine (Experimental): Intramuscular injection of 100 μg of 763SIP8 protein adjuvanted with 500 μg MPLA liposomes will be administrated 4 times (day 0, week 8, week 24 and week 48).
  Interventions: Biological: 763SIP8/MPLA-5 vaccine

INTERVENTIONS:
Biological: 763SIP8/MPLA-5 vaccine — 763SIP8/MPLA-5 vaccine at day 0, week 8, week 24 and week 48.

SUMMARY:
Study to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein SOSIP v8.2 763 Vaccine, Adjuvanted with MPLA Liposomes, in Healthy, HIV-Uninfected Adults

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged between 18 and 50 years on the day of screening.
2. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
3. Willing and able to give written informed consent.
4. Willing to undergo HIV testing, risk reduction counselling and receive HIV test results, including the possibility of vaccine-induced seropositivity (VISP).
5. If female of childbearing potential, willing to use highly effective contraceptive methods or have practiced sexual abstinence from the screening visit until four months after the last vaccination.

   Highly effective contraceptive methods will include:

   oral, intravaginal or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomized partner and sexual abstinence*
6. All female volunteers who are not heterosexually active at screening, must agree to utilize a highly effective method of contraception if they become heterosexually active, as outlined above.
7. All female volunteers must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Visits and Procedures (Appendix 1).
8. All sexually active male volunteers, regardless of reproductive potential, must be willing to use a highly effective method of contraception from the day of first vaccination until at least four months after the last vaccination to avoid exposure of partners to Investigational Medicinal Product in ejaculate and to prevent conception with female partners.
9. Willing to abstain from donating blood, eggs or sperm from the day of first vaccination until at least 3 months after receiving the last dose of the vaccine and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV antibody titres become undetectable.
10. Body Mass Index 18 to 49 Kg/m2 at screening. *A woman will be considered of childbearing potential, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. NOTE: Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method (LAM) are not acceptable methods of contraception. 8. If male and not sterilized, willing to avoid impregnating female partners from screening until 8 weeks after last injection.

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection (HIV Ag/Ab plus HIV RNA testing)
2. Self-reported risk for HIV exposure or STIs prior to screening, defined as:

   * Unprotected sexual intercourse with a known HIV infected person, a partner known to be at high risk for HIV infection or a casual partner (i.e., no continuing established relationship) in the last six months;
   * Engaged in sex work in the last twelve months;
   * Frequent excessive daily alcohol use or frequent binge drinking, or any use of illicit drugs in the last twelve months;
   * Self-reported history of newly-acquired syphilis, gonorrhoea, non-gonococcal urethritis, HSV-2, chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B in the last twelve months;
   * MSM or transgender persons having had unprotected anal intercourse in the last six months with either a male partner with an unknown HIV status OR a HIV positive partner with a (presumed) detectable viral load;
   * MSM or transgender persons diagnosed with a rectal STI in the last six months;
   * MSM or transgender persons who have been prescribed post-exposure prohylaxis (PEP) in the last six months
3. If female, pregnant or planning a pregnancy during the period of enrolment until four months after the last study vaccination; or lactating.
4. Any clinically relevant medical condition that is considered in the opinion of the investigator to make the volunteer unsuitable for participation in the study (under which underlying haematological disorders, auto-immune disease, immunodeficiency, gastrointestinal, hepatic and cardiopulmonary disorders). This also includes a history of malignancy in the past five years (prior to screening) or ongoing malignancy. (Note: A history of a completely excised malignancy that is considered cured is not an exclusion).
5. Psychiatric condition that compromises the safety of the volunteers and compliance with the protocol (severe depression, psychosis, history of suicide attempts, bipolar disorder, personality disorder, severe food disorder, use of antipsychotic medication).
6. History of respiratory disease requiring daily medication or any treatment of respiratory disease exacerbations in the last 5 years
7. Infectious disease in the six months before screening: acute and chronic hepatitis B infection (HbsAg-positive), hepatitis C infection (anti-HCV and HCV RNA positive), treatment for chronic hepatitis C infection in the past year, or active syphilis (positive chemiluminescence immunoassay (LIAISON XL), confirmed by positive RPR).
8. History of hyposplenia (anatomical or functional).
9. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions.) (Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience, is eligible).
10. History of hypersensitivity, generalized urticaria, angioedema or anaphylaxis and other significant reactions related to food, drugs, vaccines or pharmaceutical agents (Note: subjects with angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction can be included
11. Receipt of any vaccine within 30 days of vaccination with the Investigational Medicinal Product (14 days for seasonal influenza vaccination).
12. Receipt of blood products or blood-derived products within four months of screening.
13. Impossibility to proceed to the leukapheresis (e.g. absence of peripheral venous access).
14. Participation in another clinical trial of an Investigational Medicinal Product currently, within the previous three months or expected participation during this study. Concurrent participation in an observational study, not involving medicinal products and not requiring any blood or tissue sample collection is not an exclusion criterion.
15. Prior receipt of another investigational HIV vaccine or HIV monoclonal antibody (product). (Note: receipt of placebo in a previous HIV vaccine trial will not exclude a volunteer from participation if documentation is available.)
16. Known hypersensitivity to any component of the vaccine formulation used in this trial, or severe or multiple allergies to drugs or pharmaceutical agents.
17. Positive reaction in antinuclear antibody (ANA) screen and/or subsequent anti-dsDNA and/or anti-ENA assessment; or clinically significant immunoglobulin (IgA, IgG or IgM) values.
18. Use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or potentially cause harm to the volunteer. Use of corticosteroids, immunosuppressants, chemotherapeutics, anti- tuberculosis or other medications considered significant by the investigator within the previous six months. The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis (except for steroids applied to the non-dominant upper arm); or a short course (duration of ten days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least two weeks prior to enrolment in this study.
19. Active, serious infections requiring (par)enteral antibiotic, antiviral or antifungal therapy within 30 days prior to enrolment.
20. Seizure disorder: A participant who has had a seizure in the last three years prior to screening is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for three years).
21. Any of the following abnormal laboratory parameters:

    * Absolute neutrophil count ≤1,000/mm3
    * Absolute lymphocyte count ≤650/mm3
    * Hemoglobin <11 g/dl in females; <13 g/dl in males
    * Platelets < 125,000 cells/mm3
    * ALT >1.25 x ULN
    * AST>1.25 x ULN
    * Creatinine >1.1 ULN
22. If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of volunteers with a ≥ grade 3 solicited adverse (local or systemic) | from vaccination day up to 7 days post each vaccination
  Measured by ≥ grade 3 solicited adverse
Proportion of volunteers with ≥ grade 3 and/or vaccine related unsolicited adverse events | from the day of each vaccination up to 28 days post each vaccination
  Measured by ≥ grade 3 and/or vaccine related unsolicited adverse events
Proportion of volunteers with vaccine-related serious adverse events | through study completion, an average of 2 years
  Reported as SAE

SECONDARY OUTCOMES:
Proportion of volunteers with autologous neutralizing antibodies induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Autologous neutralizing antibodies determined by recombinant virus assay
  (induction in more than one third of patients will be considered a positive immunogenic response.)
Serum titres of autologous neutralizing antibodies induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Serum antibody titers determined by recombinant virus assays
  (Induction above 1:100 will be considered as a significant reponse)
Proportion of volunteers with trimer binding antibody response induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Determined with ELISA
  (induction in more than one third of patients will be considered a positive immunogenic response)
Magnitude of the trimer binding antibody response induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Determined by ELISA
  (induction of binding antibodies three folds above the threshold of detection will be considered as a significant response)
Proportion of volunteers with heterologous neutralizing antibodies induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Determined by recombinant virus assay
  (The induction of neutralizing antibodies in more than one third of patients will be considered a positive immunogenic response)
Serum titres of heterologous neutralizing antibodies against a panel of six Tier 1a/b, Tier 2 virus strains induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Determined by recombinant virus assays
  (induction of antibody titers above 1:100 will be considered as a significant response)
Proportion of volunteers with induction of Env-specific B cell responses induced by the 763SIP8/MPLA-5 vaccine | 2 weeks after each immunization
  Measured as detection of B lymphocytes binding the HIV envelope
  (Induction of responses in one third of volunteers will be considered significant from an immunogenic perspective)
B cell response | 2 weeks after each immunization.
  Measured as proportion of B lymphocytes binding the HIV envelope and comparisons will be made between individuals with low, high and durable Neutralizing Antibodies titres:
  * Env-specific plasmablast repertoire sequence analysis in peripheral blood;
  * Env-specific germline and memory B cell repertoire sequence analysis in peripheral blood

OTHER OUTCOMES:
Proportion of volunteers with and magnitude of binding antibodies to other HIV-1 Env proteins. | 2 weeks after each immunization.
  Measured by neutralization titers against a broad panel of recombinant viruses carrying the evelope from different subtypes.
  (Titers above 1:64 will be considered as significant)
Frequency of HIV-1 Env specific B cells in peripheral blood. | 2 weeks after each immunization.
  Measured by the frecuency of HIV-1 Env specific B cells in peripheral blood (An increase of two fold in comparison to basal samples will be considered significant).
Frequency of HIV-1 Env specific T(fh) cells in peripheral blood. | 2 weeks after each immunization.
  Measured by the frecuency of HIV-1 Env specific T(fh) cells in peripheral blood (An increase of two fold in comparison to basal samples will be considered significant).
Characteristics of Env-specific monoclonal antibodies (IgG) from isolated memory B cells. | 2 weeks after each immunization.
  Capacity of neutralization assessed by recombinant virus assay.
Characteristics of Env-specific monoclonal antibodies (IgG) from plasmablasts (the latter sorted according to homing receptors). | 2 weeks after each immunization.
  Capacity of neutralization assessed by recombinant virus assay.
Breadth and epitope specificity of HIV-1 Env-specific polyclonal antibodies (pAb). | 2 weeks after each immunization.
  Evaluated by epitope mapping.
Transcriptional profile of innate immune responses. | 2 weeks after each immunization.
  Hetmap will be generated and compared with expression profile of immune response genes before immunization.
Transcriptional profile of adaptive immune responses. | 2 weeks after each immunization.
  Hetmap will be generated and compared with expression profile of immune response genes before immunization.
Frequency of antibody effector functions. | 2 weeks after each immunization.
  Determined by lysis of target cell lines after incubation with plasma or isolated antibodies.
Characteristics of antibody effector functions. | 2 weeks after each immunization.
  Determined by lysis of target cell lines after incubation with plasma or isolated antibodies.
Frequency of CD4 and CD8 lymphocytes producing IFN-gamma, Tumor necrosis factor and Interleukin-2 after stimulation with HIV-envelope peptides. | 24 hours and 2 weeks after each immunization.
  Determined by AIM labelling and intracellular staining of peripheral blood lymphocytes by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain